CLINICAL TRIAL: NCT04350034
Title: Xbox Kinect™ to Promote Physical Fitness and Lean Mass in Severely Burned Children: A Randomized Controlled Trial
Brief Title: Xbox Kinect Promote Physical Fitness and Lean Mass in Severely Burned Children
Acronym: XboxBurn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qassim University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Basha, Assistant Professor, College of Medical Rehabilitation, Qassim University, Saudi Arabia, Qassim, Buraidah. Consultant Physical Therapist, El-Sahel Teaching Hospital, General Organization for Teaching Hospitals and Institutes, Cairo, Egypt., Qassim University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 2656PT
Record Dates: First submitted 2020-04-09; First posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Burns
Keywords: lean body mass; VO2 Peak; muscle strength; Enjoyment; Severely burned children; Xbox Kinect
MeSH Terms: conditions — Burns | interventions — Control Groups; Standard of Care

STUDY DESIGN:
Intervention Model Description: The Xbox group participated in a 12-week of routine physiotherapy program supplemented with Xbox training program. The control group participated in the routine physiotherapy program.
  In the study group received Xbox training, the dose of Xbox training was 50 min, three times a week for 12 weeks, using the Xbox gaming system. The games were anticipated onto a 45-inch Samsung television. The playing area was 16 * 12 m. The content of Xbox training consisted of practicing five Xbox games (Rally Ball, Reﬂex Ridge, River Rush, 2000 Leaks and parkour). Children practiced each game for 10 min, bringing about every session enduring 50 min.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xbox training group (Experimental): The study group received Xbox training plus routine physical therapy protocol treatment. The dose of Xbox training was 50 min, three times a week for 12 weeks, using the Xbox gaming system (Xbox 360 Kinect console; Microsoft Inc., Redmond, Washington, USA).
  Interventions: Other: Xbox training; Other: Control group
- Control group (Placebo Comparator): patients participated in a routine physical therapy protocol (RPTP) including joint range of motion exercises (ROM), muscle stretching technique, splinting, daily walking, and ADL training.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Xbox training — patients in this group received routine physical therapy protocol plus Xbox training.
  Before the intervention started, the Xbox group was given a 45 min introductory session on how to use the xbox adventure games and its tools. All sessions were led by a single experienced physiotherapist (different to the physiotherapist who performed the assessments tests) in order to provide instruction on how to perform each exercise.
  Other Names: interactive video games
  Arms: Xbox training group
Other: Control group — routine physical therapy protocol (RPTP) including joint range of motion exercises (ROM), muscle stretching technique, splinting, daily walking, and ADL training.
  Other Names: Standard of care

SUMMARY:
The outcome measures included quadriceps muscle strength as measured using an isokinetic dynamometer, LBM is measured by DEXA and cardiopulmonary fitness was assessed by measuring VO2 peak during a standardized treadmill exercise test using the modified Bruce protocol. All outcome measures were evaluated immediately after discharge as baseline and after 12 weeks of intervention.

DETAILED DESCRIPTION:
Forty healed pediatric burn patients (24 boys and 16 girls), aged 10 - 15 years, were enrolled from the outpatient clinic in the faculty of physical therapy, Cairo university, Egypt. The inclusion criteria were: total body surface area (TBSA) of 40-60%, being ambulatory without an assistant. The exclusion criteria included metabolic disorders, neuropathy, visual or vestibular disorders, amputation, participation in another study, any adverse medication reactions, history of epilepsy, loss of balance, and lower or upper limb deformity. All patients received similar standard medical care and treatment from the time of admission until the time of discharge.

Total burn surface area was assessed by the "modified Lund and Browder charts" method during excisional surgery immediately following hospital admittance. Informed written consent was obtained from each patient's guardian prior to enrollment.

All procedures were approved by the ethical committee of the faculty of physical therapy, Cairo university, Giza, Egypt. After consent was obtained, patients were randomly assigned to standard of care group (SOC) or Xbox training group (Xbox).

The Xbox group participated in a 12-week of routine physiotherapy program supplemented with Xbox training program (N=20). In contrast, the SOC group participated in the routine physiotherapy program (N=20).

A normal activity of daily living (ADL), diet and patient's lifestyle were maintained for all participants as much as possible.

ELIGIBILITY:
Inclusion Criteria:

* total body surface area (TBSA) of 40-60%.
* being ambulatory without an assistant.

Exclusion Criteria:

* metabolic disorders.neuropathy.
* visual or vestibular disorders.
* amputation.
* participation in another study.
* history of epilepsy.
* loss of balance.
* lower or upper limb deformity.

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-20 (Actual)

PRIMARY OUTCOMES:
VO2 peak | pre-intervention (1 month after burn injury)
  determined using a Graded Exercise Test (GXT) using a modified Bruce protocol treadmill test.
VO2 peak | after 12 weeks of treatment
  determined using a Graded Exercise Test (GXT) using a modified Bruce protocol treadmill test.

SECONDARY OUTCOMES:
Isokinetic testing Muscle strength | pre-intervention (1 month after burn injury)
  assessed using a Biodex dynamometer (Biodex Medical System, Shirley, NY,USA ).
Isokinetic testing Muscle strength | after 12 weeks of treatment
  assessed using a Biodex dynamometer (Biodex Medical System, Shirley, NY,USA ).

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated during and/or analyzed during the current study are available from the corresponding author on reasonable request.
Supporting Information: Study Protocol
Time Frame: 6 months after publication
Access Criteria: IPD will be available upon reasonable request by email from the main author after revising the requester qualification relevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] Herndon DN, Rodriguez NA, Diaz EC, Hegde S, Jennings K, Mlcak RP, Suri JS, Lee JO, Williams FN, Meyer W, Suman OE, Barrow RE, Jeschke MG, Finnerty CC. Long-term propranolol use in severely burned pediatric patients: a randomized controlled study. Ann Surg. 2012 Sep;256(3):402-11. doi: 10.1097/SLA.0b013e318265427e. PMID 22895351
- [Background] Hettiaratchy S, Papini R. Initial management of a major burn: II--assessment and resuscitation. BMJ. 2004 Jul 10;329(7457):101-3. doi: 10.1136/bmj.329.7457.101. No abstract available. PMID 15242917
- [Background] Przkora R, Herndon DN, Suman OE. The effects of oxandrolone and exercise on muscle mass and function in children with severe burns. Pediatrics. 2007 Jan;119(1):e109-16. doi: 10.1542/peds.2006-1548. Epub 2006 Nov 27. PMID 17130281
- [Derived] Basha MA, Aboelnour NH, Aly SM, Kamel FAH. Impact of Kinect-based virtual reality training on physical fitness and quality of life in severely burned children: A monocentric randomized controlled trial. Ann Phys Rehabil Med. 2022 Jan;65(1):101471. doi: 10.1016/j.rehab.2020.101471. Epub 2021 Nov 23. PMID 33316436

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-04): https://cdn.clinicaltrials.gov/large-docs/34/NCT04350034/Prot_SAP_000.pdf